CLINICAL TRIAL: NCT06329245
Title: Development of Prosocial Behaviors and Related Brain Network in Infants of High and Low Risk of ASD
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: ShanghaiTech University (Other)
Responsible Party: Sponsor
Other Study IDs: brainpro2022
Record Dates: First submitted 2024-03-19; First posted 2024-03-25 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Autism or Autistic Traits; Healthy
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high-risk group: Subjects in the case group have one or more older siblings with ASD.
  Interventions: Other: Do not take any interventions
- low-risk group: Subjects in the controlled group do not have older siblings with ASD.
  Interventions: Other: Do not take any interventions

INTERVENTIONS:
Other: Do not take any interventions — Do not take any interventions

SUMMARY:
The goal of this observational study is to compare the developmental trajectories of prosocial behaviors and functional network connections in infants and toddlers at high and low risk of autism spectrum disorder (ASD). The main questions it aims to answer are what the differences in prosocial behaviors and related brain network connections between infants/toddlers at high and low risk of ASD are. Participants will receive developmental and social communicational assessments (Griffiths Mental Developmental Scales, Peabody Developmental Motor Scales, The Communication and Symbolic Behavior Scales Developmental Profile Infant-Toddler Checklist), resting-state EEG and MRI in a natural sleeping state.

DETAILED DESCRIPTION:
The longitude observational study will be performed to compare the developmental trajectories of prosocial behaviors and functional network connections in infants and toddlers at high and low risk of autism spectrum disorder (ASD). We will follow up the subjects at 3-, 6-, 9-, 12-, 18-, 24-, 30-, and 36-month-old. Clinical diagnosis will be made on 24-month-old or after, with the DSM-5 as the diagnostic criterion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were enrolled as high-risk if they had an older sibling with a clinical diagnosis of ASD confirmed on the Autism Diagnostic Observation Schedule, second edition (ADOS-2) or Autism Diagnostic Interview (ADI-R).
* Subjects were enrolled in the low-risk group if they had an older sibling without evidence of ASD and no family history of a first or second-degree relative with ASD.

Exclusion Criteria:

1. diagnosis or physical signs strongly suggestive of a genetic condition or syndrome (e.g., fragile X syndrome) reported to be associated with ASDs;
2. a significant medical or neurological condition affecting growth, development or cognition (e.g., CNS infection, seizure disorder, congenital heart disease);
3. sensory impairment such as vision or hearing loss;
4. low birth weight (<2000 grams) or prematurity (<37 weeks gestation);
5. possible perinatal brain injury from exposure to in-utero exogenous compounds reported to likely affect the brain adversely in at least some individuals (e.g., alcohol, selected prescription medications);
6. contraindication for MRI (e.g., metal implants);
7. a family history of intellectual disability, psychosis, schizophrenia or bipolar disorder in a first-degree relative.

Ages: 0 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The longitude study will be performed in high-risk infants of ASD who have at least one older sibling with a clinical diagnosis of ASD. The low-risk group will also be recruited from healthy infants as control group if they had an older sibling without evidence of ASD and no family history of a first or second-degree relative with ASD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
clinical diagnosis | At about 2.5 to 3 year-old.
  Clinicians will diagnose subjects as ASD, other neurodevelopmental disorders, or typical developing children, using DSM-5 and ADOS-2.
neurodevelopmental outcome | At 6, 12, 18, 24, and 36-month-old.
  The neurodevelopmental outcome will be measured by Griffiths Mental Developemental Scales. The developmental ages (DA) are referred from the norms and developmental quotients (DQs) are calculated by DA/CA (chronological age)*100. Higher DQ indicates better development. The normal range of the DQ is above 70.
Prosocial behaviors | At 6, 12, 18, 24, and 36-month-old.
  The prosocial behaviors will be measured by different behavior paradigms including helper-and-hinder, crying baby, and Theory of Mind.
nuclear magnetic resonance imaging(MRI) | At 6, 12, 18, 24, and 36-month-old.
  Cranial MRI data will be collected during subjects are in natural asleep or awake, using uMR 890 3T of United Imaging company.
Event related potentials (ERPs) | At 6, 12, 18, 24, and 36-month-old.
  ERPs will be tested using eego™ mylab of ANT Neuro company. Mu suppression、N1/N2、P3/LPP will be compared between children with ASD and typical development.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Xu, doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No